CLINICAL TRIAL: NCT02601339
Title: Beside Monitor of Cerebral Metabolism in Premature Infants With Intraventricular Hemorrhage and Post-Hemorrhagic Hydrocephalus
Brief Title: NIRS Monitoring in Premature Infants
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Pei-Yi Lin, Assistant Professor, Boston Children's Hospital
Other Study IDs: 2014P001713; 1K99HD083512-01 (NIH); P00014042 (Other: Boston Children's Hospital)
Record Dates: First submitted 2015-11-06; First posted 2015-11-10 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Hemorrhage; Premature Infants; Newborn; Hydrocephalus
Keywords: spectroscopy, Near-Infrared
MeSH Terms: conditions — Hemorrhage; Premature Birth; Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- GM-IVH: Premature infants who developed germinal matrix-intraventricular hemorrhage. FDNIRS-DCS measures will be performed up to once a day if clinically feasible.
- Posthemorrhagic hydrocephalus (PHH): Premature infants with complications of hydrocephalus secondary to intraventricular hemorrhage and have the potential to receive endoscopic third ventriculostomy (ETV) with choroid plexus cauterization (CPC) and/or ventriculoperitoneal (VP) shunting for clinical treatment.
  FDNIRS-DCS measures will be performed up to once a day if clinically feasible. Additional FDNIRS-DCS measures will be performed on the day of hydrocephalus treatment to monitor the treatment response if clinically feasible. These additional measures are limited to up to four times a day.
  Interventions: Procedure: ETV/CPC
- Healthy Control (HC): Premature infants without diagnosed brain injuries. FDNIRS-DCS measures will be performed up to once a day if clinically feasible.
- Ventriculomegaly Control (VC): Infants who have symptomatic hydrocephalus of any etiology except post-hemorrhagic etiology and have the potential to receive ETV/CPC and/or VP shunting for clinical treatment.
  FDNIRS-DCS measures will be performed up to once a day if clinically feasible. Additional FDNIRS-DCS measures will be performed on the day of hydrocephalus treatment to monitor the treatment response if clinically feasible. These additional measures are limited to up to four times a day.
  Interventions: Procedure: ETV/CPC

INTERVENTIONS:
Procedure: ETV/CPC — endoscopic third ventriculostomy (ETV) combined with choroid plexus cauterization (CPC) is a surgical procedure to treat infant hydrocephalus
  Groups: Posthemorrhagic hydrocephalus (PHH); Ventriculomegaly Control (VC)

SUMMARY:
This study uses frequency domain near-infrared spectroscopy coupled with diffuse correlation spectroscopy (FDNIRS-DCS) technology for monitoring cerebral blood flow (CBF) and cerebral oxygen metabolism (CMRO2) at the bedside for newborns with germinal matrix-intraventricular hemorrhage (GM-IVH) and/or post-hemorrhagic hydrocephalus (PHH) in comparison to newborns with hydrocephalus of a different etiology (VC) and healthy controls (HC). We hypothesize that baseline cerebral metabolic dysfunction is a better biomarker for GM-IVH and PHH severity and response to PHH treatment.

This is a Boston Children's Hospital (BCH)-institutional review board(IRB) approved, multi-site study that includes collaboration with Brigham and Women's Hospital (BWH) and Beth Israel Deaconess Medical Center (BIDMC). Pei-Yi Lin receives funding from The National Institute of Health (NIH) to support the study and is the overall principal Investigator (PI) overseeing the study.

DETAILED DESCRIPTION:
Introduction and specific aims:

Germinal matrix-intraventricular hemorrhage (GM-IVH) occurs in 45% of extremely low birth weight (ELBW) premature infants, often leading to long-term neurodevelopmental impairments (NDI). Post-hemorrhagic hydrocephalus (PHH) is a common complication of GM-IVH and increases the risk of major NDI to 75-90%. Currently, the only bedside tool to assess for hemorrhage and monitor for secondary hydrocephalus is ultrasound. Although increasing ventricular size is currently used to determine need for intervention, measures based on cerebral physiology are needed to better determine the impact of the expanding ventricles on individual cerebral metabolism.

Our group has developed advanced FDNIRS-DCS technology for monitoring cerebral oxygen metabolism (CMRO2) in newborns at the bedside. We hypothesize that baseline and evoked cerebral metabolic dysfunctions are better biomarkers for GM-IVH and PHH severity and response to PHH treatment. To test our hypotheses, we will address the following specific aims:

Aim 1: Determine post-natal cerebral hemodynamics and oxygen metabolism trajectories in GM-IVH and PHH neonates with respect to normal controls and differences between PHH infants and infants affected by hydrocephalus due to other pathologies.

We hypothesize that:

1. Infants with GM-IVH have lower CBF and CMRO2 than healthy controls and the decrease is in proportion to the severity of GM-IVH. (GM-IVH vs HC)
2. Infants with PHH have lower CBF and CMRO2 than healthy controls. (PHH vs HC)
3. For infants who developed PHH, the decrease of CBF and CMRO2 is affected by both hemorrhages and the severity of hydrocephalus. (PHH vs VC)

Aim 2: Test the efficacy of cerebral hemodynamics and metabolism in detecting hydrocephalus treatment response in both PHH and VC groups.

We hypothesize that CBF and CMRO2 increase in response to treatment-associated improvements in hydrocephalus but remain depressed when response to treatment is inadequate.

Aim 3: Test the sensitivity of FDNIRS-DCS measured cerebral hemodynamics and oxygen metabolism in predicting developmental outcomes in infants with GM-IVH and PHH. We will assess neurodevelopmental outcomes in all enrolled infants at 5-7, 10-12, and 22-24 months corrected age and correlate with FDNIRS-DCS measurements of CBF and CMRO2, and related quantities with neurodevelopmental outcomes at approximately 5-7, 10-12, and 22-24 months corrected age.

ELIGIBILITY:
1. GM-IVH group:

   Inclusion criteria for GM-IVH group: born at gestational age (GA) 24-32 weeks; < 3 months old corrected-GA (cGA) at first measure or eligible for measurement within 12 weeks after the infant reaches 40 weeks post-menstrual age (PMA). Grade I-III IVH diagnosed by clinical cranial ultrasound or magnetic resonance imaging (MRI).

   Exclusion criteria for GM-IVH group: chromosomal abnormalities known at the time of enrollment; known or suspected metabolic disorder or neoplasm; critical congenital heart disease; congenital hydrocephalus; brain lesions that affect cerebral brain metabolism, other than GMH-IVH; central nervous system (CNS) infection.
2. PHH group:

   Inclusion criteria for PHH group: born at gestational age (GA) 24-37 weeks < 3 months old cGA at first measure or eligible for measurement within 12 weeks after the infant reaches 40 weeks age (PMA). PHH diagnosed by clinical cranial ultrasound or MRI.

   Exclusion criteria for PHH group: chromosomal abnormalities known at the time of enrollment; known or suspected metabolic disorder or neoplasm; critical congenital heart disease; congenital hydrocephalus; brain lesions that affect cerebral brain metabolism, other than IVH-PHH; CNS infection. Implanted devices or other devices that preclude the use of MRI.
3. HC group:

   Inclusion criteria for HC group: born at gestational age (GA) 24-32 weeks; < 3 months old cGA at first measure or eligible for measurement within 12 weeks after the infant reaches 40 weeks age (PMA); Apgar >7 at 5 min.

   Exclusion criteria for HC group: any clinical indication of brain injury or congenital brain malformation; chromosomal abnormality known at the time of enrollment; known or suspected metabolic disorder or neoplasm; critical congenital heart disease; CNS infection.
4. VC group:

Inclusion criteria for VC group: < 12 months old cGA at first measure or eligible for measurement within 1 year after the infant reaches 40 weeks age (PMA). Symptomatic hydrocephalus of any etiology or at high risk of developing hydrocephalus of any etiology, except post-hemorrhagic etiology; characterized by abnormal rate of head growth and full anterior fontanelle. Ventricular enlargement diagnosed by ultrasonography or MRI; no signs of IVH.

Exclusion criteria for VC group: known or suspected metabolic disorder or neoplasm; critical congenital heart disease; CNS infection. Implanted devices or other devices that preclude the use of MRI.

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The subject population will include premature and full-term neonates that fit criteria for one of the GM-IVH, PHH, HC, or VC groups.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
CMRO2 | 0-2 years old
  The primary outcomes are FDNIRS-DCS-measured CMRO2 trajectory.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yi Lin, PhD, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Background] Fantini S. Frequency-domain multichannel optical detector for noninvasive tissue spectroscopy and oximetry. Optical Engineering 34(1):32, 1995.
- [Background] Boas DA, Campbell LE, Yodh AG. Scattering and Imaging with Diffusing Temporal Field Correlations. Phys Rev Lett. 1995 Aug 28;75(9):1855-1858. doi: 10.1103/PhysRevLett.75.1855. No abstract available. PMID 10060408
- [Background] Wilson-Costello D, Friedman H, Minich N, Fanaroff AA, Hack M. Improved survival rates with increased neurodevelopmental disability for extremely low birth weight infants in the 1990s. Pediatrics. 2005 Apr;115(4):997-1003. doi: 10.1542/peds.2004-0221. PMID 15805376
- [Background] Roche-Labarbe N, Carp SA, Surova A, Patel M, Boas DA, Grant PE, Franceschini MA. Noninvasive optical measures of CBV, StO(2), CBF index, and rCMRO(2) in human premature neonates' brains in the first six weeks of life. Hum Brain Mapp. 2010 Mar;31(3):341-52. doi: 10.1002/hbm.20868. PMID 19650140
- [Background] Berghella V. Preterm Birth [Internet]. John Wiley & Sons; 2010. 1 p.
- [Background] Horbar JD, Carpenter JH, Badger GJ, Kenny MJ, Soll RF, Morrow KA, Buzas JS. Mortality and neonatal morbidity among infants 501 to 1500 grams from 2000 to 2009. Pediatrics. 2012 Jun;129(6):1019-26. doi: 10.1542/peds.2011-3028. Epub 2012 May 21. PMID 22614775
- [Background] Bates D, Maechler M, Bolker B, Walker S, editors. me4: Linear mixed-effects models using Eigen and S4 [Internet]. [cited 2015 Jun 2].
- [Background] Volpe JJ. Neurology of the Newborn. Elsevier Health Sciences; 2008. 1 p.
- [Background] Volpe JJ. Brain injury in premature infants: a complex amalgam of destructive and developmental disturbances. Lancet Neurol. 2009 Jan;8(1):110-24. doi: 10.1016/S1474-4422(08)70294-1. PMID 19081519
- [Background] Del Bigio MR. Cell proliferation in human ganglionic eminence and suppression after prematurity-associated haemorrhage. Brain. 2011 May;134(Pt 5):1344-61. doi: 10.1093/brain/awr052. Epub 2011 Apr 7. PMID 21478186
- [Background] Fantini S, Franceschini MA, Fishkin JB, Barbieri B, Gratton E. Quantitative determination of the absorption spectra of chromophores in strongly scattering media: a light-emitting-diode based technique. Appl Opt. 1994 Aug 1;33(22):5204-13. doi: 10.1364/AO.33.005204. PMID 20935909
- [Background] Lin PY, Roche-Labarbe N, Dehaes M, Carp S, Fenoglio A, Barbieri B, Hagan K, Grant PE, Franceschini MA. Non-invasive optical measurement of cerebral metabolism and hemodynamics in infants. J Vis Exp. 2013 Mar 14;(73):e4379. doi: 10.3791/4379. PMID 23524854